CLINICAL TRIAL: NCT07403071
Title: A Study Combining Big Data Mining With Experimental and Clinical Research to Validate the Alleviating Effect of Fish Oil on Bortezomib-Induced Peripheral Neuropathy
Brief Title: Validating Fish Oil's Role in Alleviating Bortezomib-Induced Neuropathy: A Multi-Method Study Integrating Big Data, Experimental, and Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-218-01
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Peripheral Neuropathy Due to Chemotherapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Fish Oils

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months

GROUPS / COHORTS (1):
- Multiple myeloma patients with bortezomib-induced peripheral neuropathy who are receiving oral fish
  Interventions: Dietary Supplement: Fish Oil (Containing Omega-3 Acids)

INTERVENTIONS:
Dietary Supplement: Fish Oil (Containing Omega-3 Acids) — The patients were followed up every two months to assess whether they subjectively felt an alleviation of peripheral neuropathy. The severity of peripheral neuropathy was objectively evaluated using the CTCAE criteria and the EORTC QLQ-CIPN20 scale.

SUMMARY:
The goal of this study is to find out if taking fish oil by mouth can help prevent or lessen a side effect called peripheral neuropathy in patients who are being treated with the chemotherapy drug bortezomib.

We are mainly looking to answer one question: Can fish oil reduce the chances of getting this nerve damage, or make it less severe, for these patients?

DETAILED DESCRIPTION:
* To understand the incidence of bortezomib-induced peripheral neuropathy (PN) and the resulting rates of treatment discontinuation and dose reduction, a real-world retrospective study will be conducted.

  * Potential preventive drugs for bortezomib-induced PN will be identified by mining the FDA Adverse Event Reporting System (FAERS) database.

    * The preventive effects of the candidate drugs against bortezomib-induced PN will be validated through in vivo and in vitro experiments.

      * A prospective, randomized controlled trial will be performed to confirm the efficacy of the candidate drugs in preventing bortezomib-induced PN.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 18 years or older, regardless of gender. (2) Diagnosed with multiple myeloma (MM) according to the "Guidelines for the Diagnosis and Management of Multiple Myeloma," and scheduled to receive bortezomib as first-line therapy.

  (3) Absence of baseline peripheral neuropathy prior to the initiation of bortezomib treatment.

  (4) Provision of signed informed consent.

Exclusion Criteria:

* (1) Patients with poor medication adherence. (2) Women who are pregnant or lactating. (3) Cases deemed ineligible by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had no baseline peripheral neuropathy before bortezomib treatment, developed peripheral neuropathy following bortezomib therapy, and subsequently received fish oil.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Grading of Peripheral Neuropathy according to NCI-CTCAE criteria | From enrollment to the end of treatment at 24 weeks